CLINICAL TRIAL: NCT03459937
Title: Integration of Yoga and Mindfulness for the Treatment of Obesity in Adults
Brief Title: Integration of Yoga for the Treatment of Obesity in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34AT009361 (NIH); R34AT009361 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Physical Activity; Weight Loss; Weight Change, Body
Keywords: obesity; yoga; mindfulness; weight loss; physical activity
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two intervention conditions, with assessments occurring at pre-intervention and post-intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessors will be masked to intervention condition. Selected investigators who are overseeing the intervention will also be masked to study outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha Yoga Intervention (Experimental): This intervention will be a behavioral weight loss intervention that includes group intervention session, prescribed dietary recommendations, and inclusion of Hatha Yoga.
  Interventions: Behavioral: Hatha Yoga Intervention
- Vinyasa Yoga Intervention (Experimental): This intervention will be a behavioral weight loss intervention that includes group intervention session, prescribed dietary recommendations, and inclusion of Vinyasa Yoga.
  Interventions: Behavioral: Vinyasa Yoga Intervention

INTERVENTIONS:
Behavioral: Hatha Yoga Intervention — Hatha Yoga will focus on a restorative style of Hatha yoga. Total duration will begin at 100 minutes per week and will gradually progress in 4-week intervals until achieving the prescribed dose of 300 min/wk (5 days per week for 60 minutes per day). While attending the behavioral group sessions the participants will also engage in a supervised yoga session with a trained yoga instructor. To facilitate the additional 4 days of unsupervised yoga, we will provide yoga videos that mimic the asanas (poses) and flow patterns that are taught in the supervised yoga sessions. The intervention includes prescribed dietary recommendations based on the participants' baseline body weight, and self-monitoring diaries, meal plans, and sample recipes will be provided. Intervention lessons will also include information related to behavior strategies for achieving the recommended calorie and fat intake goals. Participants will also be provided weekly group intervention sessions across the study period.
  Arms: Hatha Yoga Intervention
Behavioral: Vinyasa Yoga Intervention — Vinyasa Yoga will focus on a more vigorous form of yoga. Total duration will begin at 100 minutes per week and will gradually progress in 4-week intervals until achieving the prescribed dose of 300 min/wk (5 days per week for 60 minutes per day). While attending the behavioral group sessions the participants will also engage in a supervised yoga session with a trained yoga instructor. To facilitate the additional 4 days of unsupervised yoga, we will provide yoga videos that mimic the asanas (poses) and flow patterns that are taught in the supervised yoga sessions. The intervention includes prescribed dietary recommendations based on the participants' baseline body weight, and self-monitoring diaries, meal plans, and sample recipes will be provided. Intervention lessons will also include information related to behavior strategies for achieving the recommended calorie and fat intake goals. Participants will also be provided weekly group intervention sessions across the study period.
  Arms: Vinyasa Yoga Intervention

SUMMARY:
The focus of this study is to examine the feasibility of integrating Vinyasa yoga into a Standard Behavioral Weight Loss Intervention, to examine whether engagement differs between Vinyasa yoga and a restorative form of Hatha yoga within a Standard Behavioral Weight Loss Intervention, and to use this information to inform an expanded study to directly test the effectiveness of these interventions on weight loss in adults.

DETAILED DESCRIPTION:
The focus of this study is to examine the feasibility of integrating Vinyasa yoga into a Standard Behavioral Weight Loss Intervention, to examine whether engagement differs between Vinyasa yoga and a restorative form of Hatha yoga within a Standard Behavioral Weight Loss Intervention, and to use this information to inform an expanded study to directly test the effectiveness of these interventions on weight loss in adults. Thus, study will pursing the following aims:

* Vinyasa yoga will be integrated into the Standard Behavioral Weight Loss Intervention. This will require refinement of the Vinyasa yoga intervention to assure that this is appropriate for adults with obesity and to develop the necessary Vinyasa yoga intervention materials.
* The feasibility of randomizing and retaining participants within the context of a Standard Behavioral Weight Loss Intervention that also includes either a restorative Hatha style of yoga or Vinyasa style of yoga will be examined.
* The fidelity and compliance to the yoga components of the intervention will be examined.

To examine the aims listed above potential participants will be recruited through a variety of advertisement methods. Those individuals responding to these advertisements will have the study explained to them and informed consent will be obtained. These participants will complete a series of screening assessments that will be used to determine eligibility (height and weight to determine body mass index, resting blood pressure, heart rate, cardiorespiratory fitness). For participants deemed to be eligible and randomized to participate in this study, these measures will also be used as their baseline data from analysis. Additional data collection will be collected at the baseline assessment visit, with assessments repeated following the 6 month intervention. Assessments will include the following:

* Height and Weight
* Resting Blood Pressure and Heart Rate
* Cardiorespiratory Fitness
* Anthropometric Measures (girth of waist and hips)
* Physical Activity
* Dietary Intake
* Additional Questionnaires to assess demographics, physical activity barriers, eating behaviors, sedentary behavior, physical activity self-efficacy, mindfulness, psychological flexibility and self-regulation, affect, perceived stress, anxiety, sleep, depressive symptoms, and treatment satisfaction.

Assessments will be completed at both baseline and following the 6-month intervention. Moreover, following the intervention, participants will engage in group-based qualitative interviews. These qualitative interviews will focus on better understanding strengths, weaknesses, and barriers to engagement in the intervention that was used in this study. This information will be used to refine our approach prior to pursuing additional studies in this areas of research.

This study involves a 6 month behavioral weight loss intervention (SBWI) with participants randomized to either Hatha Yoga or Vinyasa Yoga as the form of physical activity. All randomized participant will received the components of the SBWI along with either Hatha Yoga or Vinyasa Yoga based on their randomized intervention assignment. Participants will attend weekly group meetings for all weeks of the study. Group meetings will last approximately 30-45 minutes in duration and will be led by trained behavioral interventionists with previous experience facilitating behavioral weight loss intervention meetings. These meetings will focus on strategies to promote behavior change and weight management. Strategies to promote behavior change will included the Social Cognitive Theory, Problem Solving Theory, and Relapse Prevention. Participants will be weighed weekly prior to group meetings to track changes in weight throughout the study and assist interventionists with weight counseling. Participants who do not attend the weekly group meeting will be contacted via telephone call to reschedule for an individual weigh-in and make-up session with an interventionist prior to the next group meeting. If an individual make-up session cannot be scheduled, an interventionist will provide a brief counseling session by telephone and the written materials will be mailed to the participant.

Dietary recommendations within the intervention will be based on the participants' baseline body weight. These calorie goals are based on intake recommendations that have been successful in other weight loss programs, and fat intake goals are consistent with the USDA Dietary Guidelines. Participants weighing less than 200 pounds will be prescribed a 1200 kcal/day diet, participants weighing between 200 to less than 250 will be prescribed 1500 kcal/day, and participants weighing 250 or more will be prescribed 1800 kcal/day. To promote adoption and adherence to these recommendations, participants will be provided self-monitoring paper diaries, meal plans, and sample recipes. Participants will be instructed to self-monitor daily and will be instructed to turn in self-monitoring food diaries to their interventionist prior to group intervention meetings. Printed intervention lessons will also include information related to behavior strategies for achieving the recommended calorie and fat intake goals.

Physical Activity Components of the Intervention:

Hatha Yoga Group: The specific description of physical activity for those randomized to receive Hatha Yoga will focus on a restorative style of Hatha yoga. This will involve a systematic progression to allow for participants to acclimate to the poses and this style of yoga practice. Total duration will begin at 100 minutes per week and will gradually progress in 4-week intervals until achieving the prescribed dose of 300 min/wk (5 days per week for 60 minutes per day). Participants will be instructed to spread this dose of activity equally across 5 days each week, with each session starting at 20 minutes and progressing to 50 minutes. The initial 1-2 weeks will focus on the participants understanding the asanas (or poses) and gaining kinesthetic awareness of their body while moving through the movement sequences. Study participants will be provided with a yoga mat to use throughout the study, and they will be permitted to keep this yoga mat at the conclusion of their participation in this study.

While attending the SBWI group session the participants will also engage in a supervised yoga session with a trained yoga instructor. To facilitate the additional 4 days of unsupervised yoga, yoga videos that we develop that mimic the asanas (poses) and flow patterns that are taught in the supervised yoga sessions will be provided, and these videos will be led by the same individual who is instructing the supervised yoga sessions. To facilitate the use of these yoga videos by participants, access will be provided by loading them on to a tablet (iPad, Surface, etc.) that will be provided to the participant or through other electronic formats (YouTube Channel, streaming through study website, etc.). The sequence of videos will be scheduled to be accessible to the participant on predetermined dates that coincide with the progression of the yoga activities in the intervention.

Vinyasa Yoga Group: The specific description of physical activity for those randomized to receive Vinyasa Yoga will focus on a more vigorous form of yoga. This will involve a systematic progression to allow for participants to acclimate to the poses and this style of yoga practice. Total duration will begin at 100 minutes per week and will gradually progress in 4-week intervals until achieving the prescribed dose of 300 min/wk (5 days per week for 60 minutes per day). Participants will be instructed to spread this dose of activity equally across 5 days each week, with each session starting at 20 minutes and progressing to 50 minutes. The initial 1-2 weeks will focus on the participants understanding the asanas (or poses) and gaining kinesthetic awareness of their body while moving through the movement sequences. Study participants will be provided with a yoga mat to use throughout the study, and they will be permitted to keep this yoga mat at the conclusion of their participation in this study.

While attending the SBWI group session the participants will also engage in a supervised yoga session with a trained yoga instructor. To facilitate the additional 4 days of unsupervised yoga, yoga videos that we develop that mimic the asanas (poses) and flow patterns that are taught in the supervised yoga sessions will be provided, and these videos will be led by the same individual who is instructing the supervised yoga sessions. To facilitate the use of these yoga videos by participants, access will be provided by loading them on to a tablet (iPad, Surface, etc.) that will be provided to the participant or through other electronic formats (YouTube Channel, streaming through study website, etc.). The sequence of videos will be scheduled to be accessible to the participant on predetermined dates that coincide with the progression of the yoga activities in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females of all race/ethnic groups are eligible for participation in this study.
* 18-60 years of age.
* Body mass index (BMI) between 25.0 to <40.0 kg/m2.
* Ability to provide informed consent prior to participation in this study.
* Ability to provide clearance from their primary care physician to engage in the diet and physical activity components of the weight loss intervention.

Exclusion Criteria:

* Report moderate-to-vigorous exercise on >3 days per week or a total of >60 minutes per week over the past 3 months.
* Engaging in any style of yoga on an average of at least 1 day per week over the past 3 months.
* Report weight loss of >3% or participating in a weight reduction diet in the past 3 months.
* Females who are pregnant or breastfeeding, or reporting a planned pregnancy during the study period.
* History of bariatric surgery.
* Report current medical condition or treatment for a medical condition that could affect body weight. These may include the following: diabetes mellitus; hyperthyroidism; inadequately controlled hypothyroidism; chronic renal insufficiency; chronic liver disease; cancer; gastrointestinal disorders including ulcerative colitis, Crohn's disease, or malabsorption syndromes; etc.
* Current congestive heart failure, angina, uncontrolled arrhythmia, symptoms indicative of an increased acute risk for a cardiovascular event, prior myocardial infarction, coronary artery bypass grafting or angioplasty, conditions requiring chronic anticoagulation (i.e. recent or recurrent DVT).
* Resting systolic blood pressure of >160 mmHg or resting diastolic blood pressure of >100 mmHg.
* Eating disorders that would contraindicate weight loss or physical activity.
* Alcohol or substance abuse.
* Currently treated for psychological issues (i.e., depression, bipolar disorder, etc.), taking psychotropic medications within the previous 12 months, or hospitalized for depression within the previous 5 years.
* Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance at scheduled intervention sessions or assessments.
* Physical activity or weight loss deemed to be contraindicated based on response to the cardiorespiratory fitness test that will be conducted as part of the screening procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Fidelity to the yoga interventions | Across the 6 month intervention period
  Fidelity will be based on the number of days that yoga was performed during the intervention compared to the prescribed number of days that yoga was to be completed in both the Hatha Yoga Group and the Vinyasa Yoga Group
Compliance to the yoga interventions | Across the 6 month intervention period
  Compliance will be based on the number of days that the yoga was completed at the prescribed duration compared to the prescribed number of days that yoga was to be completed in both the Hatha Yoga Group and the Vinyasa Yoga Group

OTHER OUTCOMES:
Weight | Change at 6 months
  Body weight will be assessed in kilograms
Height | Change at 6 months
  Height will be measured in centimeters
Body Mass Index (BMI) | Change at 6 months
  measures of weight and height will be combined to report BMI in kg/m2
Cardiorespiratory Fitness | Change at 6 months
  Cardiorespiratory fitness will be measured using a submaximal graded exercise test.
Physical Activity Counts | Change at 6 months
  Physical activity counts will be assessed using actigraphy.
Physical Activity minutes | Change at 6 months
  Physical activity minutes will be assessed using questionnaires.
Physical Activity Energy Expenditure | Change at 6 months
  Physical activity energy expenditure (kcal/week) will be assessed using questionnaires.
Dietary Intake | Change at 6 months
  Dietary intake (kcal/day) will be measured using a food frequency questionnaire
Sedentary Behavior Duration | Change at 6 months
  Sedentary behavior duration (minutes) will be assessed using questionnaires
Sedentary Behavior Counts | Change at 6 months
  Sedentary behavior will be assessed from counts using actigraphy
Physical activity barriers | Change at 6 months
  Physical activity barriers will be assessed with a questionnaire
Eating behaviors | Change at 6 months
  Eating behaviors will be assessed with questionnaires
Mindfulness | Change at 6 months
  Mindfulness will be assessed with questionnaires
Psychological flexibility | Change at 6 months
  Psychological flexibility will be assessed with questionnaires
Self-regulation | Change at 6 months
  Self-regulation will be assessed with questionnaires
Affect | Change at 6 months
  Affect will be assessed with a questionnaire
Depressive symptoms | Change at 6 months
  Depressive symptoms will be assessed with questionnaires
Anxiety | Change at 6 months
  Anxiety will be assessed with questionnaires
Sleep time | Change at 6 months
  Sleep time will be assessed with a questionnaire
Sleep quality | Change at 6 months
  Sleep quality will be assessed with a questionnaire
Sleep duration | Change at 6 months
  Sleep duration will be assessed with counts from actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakicic JM, Davis KK, Rogers RJ, Sherman SA, Barr S, Marcin ML, Collins KA, Collins AM, Yuan N, Lang W. Feasibility of Integration of Yoga in a Behavioral Weight-Loss Intervention: A Randomized Trial. Obesity (Silver Spring). 2021 Mar;29(3):512-520. doi: 10.1002/oby.23089. Epub 2021 Feb 2. PMID 33528905